CLINICAL TRIAL: NCT05309252
Title: The Unmet Needs and the Workplace Reintegration of Breast Cancer Patients: the NEW-BreCa Project
Acronym: NEW-BreCa
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Sara Paltrinieri, MSc Occupational Therapist, Azienda USL Reggio Emilia - IRCCS
Other Study IDs: 2022/0035983
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Cancer Survivors; Unmet needs; Supportive care needs; Return to Work; Epidemiology; Observational study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer (BC) have unmet needs that can impact negatively on participation in meaningful activities and the overall quality of life, if not addressed by the healthcare services. One of those needs is the return to work (RTW) for female in their working age.

The perceived needs of BC patients and RTW process might be influenced by sociodemographic data, disease-related, and work-related factors. Moreover, needs might change (type and priority) from diagnosis onwards. Prospective data regarding these topics have never been collected in Italian BC patients.

DETAILED DESCRIPTION:
BC accounts for one of the highest worldwide public health burden, representing a population with increasing trends in Western countries. In Italy, BC is the most common diagnosis in female sex across all age groups, and the 50% were in their working age (between 20 and 64 years old).

Although early diagnostic methods and effective treatments offer BC patients a longer lifespan, the effects of therapies negatively impact on patients' daily lives and quality of life. BC patients might perceive variable needs (e.g., information, psychological) related to the experience of cancer and the care process that are considered as necessary to achieve goals in everyday life and return to normalcy. Unmet needs may arise when a gap occurs between a person's experience of healthcare services and the actual services require. Thus, care models for this population should be planned in the light of the most recent evidences.

Although the RTW is one of the necessities of BC patients, cancer survivors are more likely to be unemployed than healthy individuals and some difficulties may occur during the RTW process. Sociodemographic data, disease-related, and work-related factors might act as predictors of the unmet needs perceived by BC patients and the employment status from diagnosis onwards.

In Italy, unmet needs and RTW of BC patients have been investigated only through cross-sectional studies.

This type of study design does not allow to determine the causal relationship between potential determinants and unmet needs and occupational status, as well as the changes occurred from the diagnosis onwards. Prospective data regarding these topics have never been collected in Italian BC patients.

Thus, the investigators aim (1) to investigate the factors that could predict job loss, work difficulties, and long-term sick leave in BC patients of working age and (2) to investigate the factors that could predict the daily life needs of BC patients.

The investigators have planned a prospective data collection that will last 24 months. During the observations, the investigators will collect sociodemographic data, disease-related, and work-related factors.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer diagnosis (regardless of stage and treatment)
* breast cancer patients in adulthood (≥ 18 years)
* breast cancer patient who will participate to an educational group session held by the physiotherapists of the PMRU

For patients who are not in working age or not employed at diagnosis, the work-related factors will not be collected.

Exclusion Criteria:

* breast cancer patients who do not speak fluently italian language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit breast cancer patients from those who will participate to an educational group session held by the physiotherapists of the Physical Medicine and Rehabilitation Unit (PMRU).
  Breast cancer patients who undergo surgery are offered to participate voluntarily in this educational group session after inpatients.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
occupational status | 12 months
  the identification of the occupational status at first contact and at the following observations. At each observation, we will ask the participants if they have returned to work or not
work difficulties | 12 months
  the collection of the work-related difficulties that will be counted and classified using the Core Set-VR-Onco and, then, described qualitatively
sick leave | 12 months
  the number of days of sick leave
perceived needs | 12 months
  the identification of the perceived needs at first contact and at the following observations

CONTACTS AND LOCATIONS:
Overall Officials: Sara Paltrinieri, Msc OT, Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Azienda Unità Sanitaria Locale Reggio Emilia, Reggio Emilia, Italy